CLINICAL TRIAL: NCT00796900
Title: Dantrolene as a Treatment for Hyperthermia in Patients After Subarachnoidal Hemorrhage
Brief Title: Dantrolene for Treatment of Hyperthermia in Subarachnoidal Hemorrhage (SAH)
Acronym: DTH1
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: organizationally not possible
Sponsor: Medical University of Vienna (Other)
Responsible Party: Andrea Holzer, MD, Medical University Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK 197/2004
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2009-09

CONDITIONS: Hyperthermia
Keywords: Hyperthermia; subarachnoidal hemorrhage; placebo controlled; double blinded; Dantrolene
MeSH Terms: conditions — Hyperthermia | interventions — Dantrolene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dantrolene (Experimental)
  Interventions: Drug: Dantrolene
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dantrolene — Patients who satisfy the inclusion/exclusion criteria of the study and who are enrolled in this study will be randomized with computer-generated grouping to either one of two groups. One group of subjects will be given dantrolene for the first episode of fever. The other group will be given placebo. Dantrolene is supplied in 70-ml vials containing 20 mg dantrolene. Dantrolene will be given in the following dose: 5 mg/kg BW given intravenously over 30 minutes. As placebo NaCl 0,9% will be used.
  Arms: Dantrolene
Drug: Placebo — Patients who satisfy the inclusion/exclusion criteria of the study and who are enrolled in this study will be randomized with computer-generated grouping to either one of two groups. One group of subjects will be given dantrolene for the first episode of fever. The other group will be given placebo. Dantrolene is supplied in 70-ml vials containing 20 mg dantrolene. Dantrolene will be given in the following dose: 5 mg/kg BW given intravenously over 30 minutes. As placebo NaCl 0,9% will be used.
  Arms: Placebo

SUMMARY:
Dantrolene is used to prevent hyperthermia in intensive care patients suffering from subarachnoidal hemorrhage.

DETAILED DESCRIPTION:
Background:

Fever episodes occur in more than 50% of patients admitted to the ICU for subarachnoidal hemorrhage, central nervous system infection, seizure control, hemorrhagic stroke, and closed head injury despite antibiotic and antipyretic therapy.

The exact mechanism of hyperthermia-induced brain injury is not known; however, various processes may be involved. For example, hyperthermia might increase the release of excitatory neurotransmitter or trigger an abundant amount of oxygen free radicals. Hyperthermia may also aggravate blood-brain barrier disruption, impair cytoskeletal proteolysis, and/or enhance inhibition of enzymatic protein kinases, which, in turn, would impair recovery of energy metabolism. Antipyretics are effective for conventional fever, but less useful for various central hyperthermia syndromes, especially those resulting from strokes, SAH, and head injuries. Even aggressive cooling is usually insufficient in patients with fever because it is unable to overcome the high metabolic rate in these patients. Likewise, physical cooling is counteracted by the thermoregulatory defenses being activated to maintain hyperthermia. In non-sedated individuals, active cooling increases metabolic stress without decreasing core temperature at all. To date, treatment of centrally mediated hyperthermia remains unsatisfying.

Dantrolene has been available since 1975 as a specific treatment for acute malignant hyperthermia crises. However, dantrolene is increasingly being used for emergency treatment of life-threatening hyperthermia that is unresponsive to conventional treatments. For example, the drug has been used with some success for acute treatment of life-threatening hyperthermia resulting from neuroleptic malignant syndrome and hyperthermia associated with overdoses of various drugs. It has also been used for treatment of various other types of hyperthermia.

Efficacy in these cases appears to be based on a non-specific action of the drug; but to the extent dantrolene is effective, its action must conform to the laws of thermodynamics. Dantrolene must, therefore, reduce metabolic heat production, augment systemic heat loss, or alter the normal distribution of heat within the body. In other words, dantrolene must reverse the abnormal (or ineffective) thermoregulatory control that initiates the hyperthermic crises.

Item:

We propose to test the hypothesis that dantrolene will reduce centrally mediated fever in patients after subarachnoidal hemorrhage. Specifically, we will test the hypothesis that dantrolene decreases the magnitude and duration of hyperthermia.

The study will be restricted to neurosurgical patients with sustained fever (≥38ºC for more than an hour) without an identifiable infectious cause after subarachnoidal hemorrhage aged from 18 to 80 years. There will be no limitation of enrollment as to patients breathing spontaneously or being ventilator dependant.

ELIGIBILITY:
Inclusion Criteria:

* neurosurgical patients after subarachnoidal hemorrhage
* breathing spontaneously or being ventilator dependant
* sustained fever (≥38ºC for more than an hour) without an identifiable infectious cause.

Exclusion Criteria:

* infection
* pregnancy
* arrhythmia
* muscular dystrophia
* acute liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Magnitude and Duration of Hyperthermia | 8 hours, every 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Holzer, MD, Principal Investigator — Medical University Vienna, Department of Anesthesiology and General Intensive Care Medicine
Locations (1):
- Medical University Vienna, Vienna, Austria